CLINICAL TRIAL: NCT05190120
Title: Effects of Ultrasound-guided Adductor Canal Block Versus Femoral Nerve Block on Pain and Quadriceps Strength After Ambulatory Knee Arthroscopic Surgery
Brief Title: Adductor Canal Block Versus Femoral Block on Pain and Quadriceps Strength
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-13071
Record Dates: First submitted 2021-11-16; First posted 2022-01-13 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament Tear; Knee Meniscus Tear
Keywords: Knee arthroscopy; ACL reconstruction; Femoral block; Adductor Canal Block
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Femoral Block (Active Comparator): Patients scheduled for knee arthroscopy will have a femoral nerve block done using 0.5% ropivacaine 20ml before surgery.
  Interventions: Procedure: Femoral Nerve Block; Drug: preoperative Femoral Nerve Block using 20ml of 0.5% ropivacaine
- Adductor Canal Block (Experimental): Patients scheduled for knee arthroscopy will have an adductor canal block done using 0.75% ropivacaine 13.3ml before surgery.
  Interventions: Procedure: Adductor Canal Nerve Block; Drug: Preoperative Adductor canal block with 0.75%% ropivacaine 13.3ml.

INTERVENTIONS:
Procedure: Femoral Nerve Block — Patients having ACL reconstruction, meniscus surgery and knee arthroscopy
  Arms: Femoral Block
Procedure: Adductor Canal Nerve Block — Patients having ACL reconstruction, meniscus surgery and knee arthroscopy
  Arms: Adductor Canal Block
Drug: preoperative Femoral Nerve Block using 20ml of 0.5% ropivacaine
  Arms: Femoral Block
Drug: Preoperative Adductor canal block with 0.75%% ropivacaine 13.3ml.
  Arms: Adductor Canal Block

SUMMARY:
The purpose of this study is to compare the effects of a femoral nerve block vs. an adductor canal block on pain and quadriceps muscle strength for knee arthroscopy surgery.

DETAILED DESCRIPTION:
Patients undergoing arthroscopic knee surgery (ACL and non-ACL surgery) typically receive an ultrasound-guided femoral nerve block or an adductor canal block in the pre-operative phase for post-operative pain control. While an effective method for post-operative analgesia, the femoral nerve block is associated with profound quadriceps weakness for the duration of the nerve block, which can impair ambulation, rehabilitation, and increase the risk of falls. The more distal adductor canal block, however, contains primarily sensory branches of the femoral nerve and has been been purported by small volunteer studies to provide equally effective analgesia with minimal motor block and quadriceps weakness (as compared to femoral nerve block).

The investigators will prospectively randomize patients undergoing knee arthroscopy at the UCSF Orthopaedic Institute to receive either a single-shot femoral nerve or adductor canal block pre-operatively after taking baseline measurements of quadriceps strength (quantified by maximum voluntary isometric contraction). The quadriceps muscle strength will be checked 20 minutes after the nerve block to assess strength. All patients will subsequently undergo a general anesthetic. The primary outcome variable will be post-block quadriceps strength as a percentage of baseline from pre-block values. Secondary outcome variables that will also investigated include: VAS pain score in the post anesthesia recovery unit and post-operative day 1, duration of nerve blockade, and perioperative opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia I-III classification,
* Scheduled for arthroscopic knee surgery (meniscal debridement/repair, ACL reconstruction)

Exclusion Criteria:

* Age younger than 18 years
* Non-English speaking
* Any contraindication for regional anesthesia, such as allergy to local anesthetics or opioids, -Coagulopaty or severe thrombocytopenia
* Infection at puncture sites
* Pre-existing neuropathy in operative limb
* Need for post-operative nerve function monitoring
* Dementia
* Patient refusal
* High pre-operative opioid requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Aleshi, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Orthopedic Trauma Service, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be shared only if required for the publication of data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Femoral Block for Knee Arthroscopy/Meniscus Surgery: Patients scheduled for knee arthroscopy will have a femoral nerve block done using 0.5% ropivacaine 20ml before surgery.
- Adductor Canal Block for Knee Arthroscopy/Meniscus Surgery: Patients scheduled for knee arthroscopy will have an adductor canal block done using 0.75% ropivacaine 13.3ml before surgery.
- Femoral Block for ACL Reconstruction: Patients scheduled for ACL reconstruction will have a sciatic nerve block and a femoral nerve block done using 0.5% ropivacaine 20ml before surgery.
- Adductor Canal Block for ACL Reconstruction: Patients scheduled for ACL reconstruction will have a sciatic nerve block and an adductor canal block done using 0.75% ropivacaine 13.3ml before surgery.
Period: Overall Study
Arm/Group | Femoral Block for Knee Arthroscopy/Meniscus Surgery | Adductor Canal Block for Knee Arthroscopy/Meniscus Surgery | Femoral Block for ACL Reconstruction | Adductor Canal Block for ACL Reconstruction
Started | 31 | 35 | 33 | 33
Completed | 25 | 34 | 30 | 27
Not Completed | 6 | 1 | 3 | 6
Not completed — Lost to follow up for primary outcome measurement d/t lack of time to complete before surgery | 1 | 1 | 1 | 3
Not completed — Lost to Follow-up | 5 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: The data collection forms were missing for 10 participants. The data are not available to report, these data do not exist.
Groups:
- Total: Total of all reporting groups
Arm/Group | Femoral Block for Knee Arthroscopy/Meniscus Surgery | Adductor Canal Block for Knee Arthroscopy/Meniscus Surgery | Femoral Block for ACL Reconstruction | Adductor Canal Block for ACL Reconstruction | Total
Number analyzed (Participants) | 26 | 35 | 31 | 30 | 122
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [33 to 54] | 49 [35 to 56] | 35 [28 to 40] | 33.5 [25 to 38] | 36.5 [29 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 14 | 14 | 46
  Male | 18 | 25 | 17 | 16 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19 | 21 | 16 | 24 | 80
  Asian | 4 | 8 | 10 | 5 | 27
  Black | 1 | 1 | 0 | 0 | 2
  Hispanic/Latino | 2 | 4 | 5 | 1 | 12
  Native American or Pacific Islander | 0 | 1 | 0 | 0 | 1
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 24.3 [22.4 to 26.6] | 28.3 [24.2 to 31.8] | 25.4 [23.5 to 27.1] | 24.4 [22.8 to 25.8] | 25.3 [23.0 to 28.1]

OUTCOME MEASURES:

1. Primary Outcome: Change in Quadriceps Strength Related to the Nerve Block
Description: Quadriceps strength will be tested with a dynamometer before the nerve block and 20 minutes after the nerve block prior to surgery. The dynamometer measures the strength of the quadriceps muscles in the seated position while pushing against the device. We are trying to measure the effect of both femoral and adductor canal nerve blocks on quadriceps strength.
Time Frame: Baseline and 20 minutes after the block prior to surgery
Population: The participants with data available are reported here.
Measure: Median (Inter-Quartile Range); unit: Newtons
Arm/Group | Femoral Block for Knee Arthroscopy/Meniscus Surgery | Adductor Canal Block for Knee Arthroscopy/Meniscus Surgery | Femoral Block for ACL Reconstruction | Adductor Canal Block for ACL Reconstruction
Number analyzed (Participants) | 25 | 34 | 27 | 24
Newtons | -0.42 [-1.2 to 0.23] | -0.55 [-1.43 to -0.067] | -3.19 [-4.25 to -1.73] | -0.77 [-1.63 to 0]

2. Secondary Outcome: Numerical Pain Score From 0-10
Description: As this is an outpatient surgery, we will collect Numerical Pain Scores from the recovery room medical record after surgery as well as from the patients for the first 24 hours after surgery by contacting them at home the following day. We will evaluate the difference in patient pain scores between the two nerve blocks under study.
  The highest pain score for the 24-hour post-op period was collected for each participant. The median is reported for all participants. A pain score of 10 represents the worst pain.
Time Frame: worse pain in first 24 hours
Population: The participants with data available are reported here.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Femoral Block for Knee Arthroscopy/Meniscus Surgery | Adductor Canal Block for Knee Arthroscopy/Meniscus Surgery | Femoral Block for ACL Reconstruction | Adductor Canal Block for ACL Reconstruction
Number analyzed (Participants) | 24 | 32 | 31 | 30
score on a scale | 4.5 [3 to 6.5] | 5 [3 to 7] | 7 [4 to 9] | 6.5 [5 to 9]

3. Secondary Outcome: Duration of Nerve Block
Description: Patients will be contacted after surgery to determine when the nerve block wore off based on their increase in pain
Time Frame: 8 to 24 hours
Population: The participants with data available are reported here.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Femoral Block for Knee Arthroscopy/Meniscus Surgery | Adductor Canal Block for Knee Arthroscopy/Meniscus Surgery | Femoral Block for ACL Reconstruction | Adductor Canal Block for ACL Reconstruction
Number analyzed (Participants) | 18 | 25 | 29 | 28
minutes | 678 [454 to 903] | 731 [566 to 896] | 889 [730 to 1048] | 923 [755 to 1091]

4. Secondary Outcome: Opioid Consumption Reported at mg of Morphine Equivalence
Description: Data on the amount of pain medication consumed for the 1st 24 hours after surgery will be collected based on medications that were administered during surgery, in the recovery room and medications that patients took at home after discharge from the recovery room. All pain medications will be converted to morphine equivalence in milligrams and reported that way. The comparison will be the difference in mg morphine equivalence consumption between the two nerve block groups.
Time Frame: 2 days
Population: The participants with data available are reported here.
Measure: Median (Inter-Quartile Range); unit: Morphine milligram equivalents (MME)
Arm/Group | Femoral Block for Knee Arthroscopy/Meniscus Surgery | Adductor Canal Block for Knee Arthroscopy/Meniscus Surgery | Femoral Block for ACL Reconstruction | Adductor Canal Block for ACL Reconstruction
Number analyzed (Participants) | 22 | 32 | 30 | 30
Morphine milligram equivalents (MME) | 40 [30 to 60] | 51.25 [40 to 70] | 20 [10 to 40] | 20 [15 to 40]

ADVERSE EVENTS:
Time Frame: Day of surgery and 24 hours post-operatively
Arm/Group | Femoral Block for Knee Arthroscopy/Meniscus Surgery | Adductor Canal Block for Knee Arthroscopy/Meniscus Surgery | Femoral Block for ACL Reconstruction | Adductor Canal Block for ACL Reconstruction
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/35 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/35 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/35 | 0/33 | 0/33

LIMITATIONS AND CAVEATS:
A longer length of study time due to periods of elapsed time without a clinical research investigator to continue and complete the study, extended length of study due to COVID-19 pandemic and inability to enroll patients for an extended period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT05190120/Prot_SAP_000.pdf